CLINICAL TRIAL: NCT01264770
Title: (OSKIRA-4): A Phase IIB, Multi-Centre, Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study of the Efficacy and Safety of Fostamatinib Disodium Monotherapy Compared With Adalimumab Monotherapy in Patients With Active Rheumatoid Arthritis
Brief Title: Evaluation of Efficacy and Safety of Fostamatinib Monotherapy Compared With Adalimumab Monotherapy in Patients With Rheumatoid Arthritis (RA)
Acronym: OSKIRA -4
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: AZ decision to discontinue fostamatinib development in RA; rights to fostamatinib returned to Rigel Pharmaceuticals.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4300C00004; 2010-023692-26 (EudraCT Number)
Record Dates: First submitted 2010-12-17; First posted 2010-12-22 (Estimated); Results first posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; OSKIRA; fostamatinib
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Dosing Group A (Experimental): Oral treatment and subcutaneous injection
  Interventions: Drug: Fostamatinib and placebo injections
- Dosing Group B (Experimental): Oral treatment and subcutaneous injection
  Interventions: Drug: Fostamatinib and placebo injections
- Dosing Group C (Experimental): Oral treatment and subcutaneous injection
  Interventions: Drug: Fostamatinib and placebo injections
- Dosing Group D (Active Comparator): Oral treatment and subcutaneous injection
  Interventions: Drug: Adalimumab and placebo of fostamatinib
- Dosing Group E (Placebo Comparator): Oral treatment and subcutaneous injection
  Interventions: Drug: Placebo of fostamatinib, fostamatinib, and placebo injections

INTERVENTIONS:
Drug: Fostamatinib and placebo injections — Fostamatinib 100mg twice daily and placebo injection once every two weeks
  Arms: Dosing Group A
Drug: Fostamatinib and placebo injections — Fostamatinib 100mg twice daily / fostamatinib 150mg once daily and placebo injection once every two weeks
  Arms: Dosing Group B
Drug: Fostamatinib and placebo injections — Fostamatinib 100mg twice daily / fostamatinib 100mg once daily and placebo injection once every two weeks.
  Arms: Dosing Group C
Drug: Adalimumab and placebo of fostamatinib — Adalimumab 40mg injection once every two weeks and placebo to fostamatinib twice daily.
  Other Names: Humira®
  Arms: Dosing Group D
Drug: Placebo of fostamatinib, fostamatinib, and placebo injections — Placebo injection once every two weeks. Placebo to fostamatinib for six weeks, followed by fostamatinib 100mg twice daily (Group F) / fostamatinib 100mg twice daily then 150mg once daily (Group G).
  Arms: Dosing Group E

SUMMARY:
The purpose of the study is to evaluate the improvements in signs and symptoms of rheumatoid arthritis (RA) for fostamatinib compared to placebo or adalimumab in patients who are Disease-Modifying anti-rheumatic drug (DMARD) naïve, DMARD intolerant or have had an inadequate response to DMARDs. The study will last for approximately six months

DETAILED DESCRIPTION:
Sub-study:

Full title: Optional Genetic Research

Date: 10 September 2010

Version: 1

Objectives: To collect and store, with appropriate consent , DNA samples for future exploratory research into genes/genetic variation that may influence response (ie, absorption, distribution, metabolism and excretion, safety, tolerability and efficacy) to fostamatinib disodium and/or adalimumab; and/or susceptibility to, progression of and prognosis of RA

The main study recruitment is complete, and sub study recruitment will continue until the target is reached, estimated to be June 2013

Sub-study:

Full title: (Sub-study to OSKIRA-4): A Phase IIB, Multi-Centre, Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study of the Efficacy and Safety of Fostamatinib Disodium Monotherapy Compared with Placebo or Adalimumab Monotherapy in Patients with Active Rheumatoid Arthritis: Magnetic Resonance Imaging Sub-Study

Date: 21 March 2011

Version: 1

Primary objective: Assess the efficacy of fostamatinib in reducing joint synovial disease activity as measured by:

* Change from baseline to Week 6 (versus placebo) in OMERACT RAMRIS synovitis score.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and over
* Active rheumatoid arthritis (RA) diagnosed after the age of 16 and diagnosis within 5 years prior to study visit 1 and inadequate response to treatment with a maximum 2 Disease-Modifying anti-rheumatic drug (DMARD) therapies, or diagnosis within 5 years prior to study visit 1 and intolerance to DMARD therapy, or diagnosis within 2 years prior to study visit 1 and no previous use of DMARDs
* 4 or more swollen joints and 4 or more tender/painful joints (from 28 joint count) and either Erythrocyte Sedimentation Rate (ESR) blood result of 28mm/h or more, or C-Reactive Protein (CRP) blood result of 10mg/L or more
* At least 2 of the following: documented history or current presence of positive rheumatoid factor (blood test), radiographic erosion within 12 months prior to study enrolment, presence of serum anti-cyclic citrullinated peptide antibodies (blood test)

Exclusion Criteria:

* Females who are pregnant or breast feeding
* Poorly controlled hypertension
* Liver disease or significant liver function test abnormalities
* Certain inflammatory conditions (other than rheumatoid arthritis), connective tissue diseases or chronic pain disorders
* Recent or significant cardiovascular disease
* Significant active or recent infection including tuberculosis
* Previously received treatment with a TNF alpha antagonist (including etanercept, certolizumab, adalimumab, infliximab, golimumab) or anakinra or previous treatment with other biological agent including rituximab, abatacept and tocilizumab
* Use of any DMARDs within 6 weeks before first study visit
* Severe renal impairment
* Neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil MacKillop, MD PhD, Study Director — AstraZeneca
Locations (105):
- United States (40):
  - Research Site, Birmingham, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Huntington Beach, California
  - Research Site, Long Beach, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Daytona Beach, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Pinellas Park, Florida
  - Research Site, Venice, Florida
  - Research Site, Chicago, Illinois
  - Research Site, South Bend, Indiana
  - Research Site, Bowling Green, Kentucky
  - Research Site, Elizabethtown, Kentucky
  - Research Site, Oxon Hill, Maryland
  - Research Site, Kalamazoo, Michigan
  - Research Site, Richmond Heights, Missouri
  - Research Site, Kalispell, Montana
  - Research Site, Nashua, New Hampshire
  - Research Site, Albuquerque, New Mexico
  - Research Site, Las Cruces, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Perrysburg, Ohio
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Jackson, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
- Bulgaria (6):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sevlievo
  - Research Site, Sofia
  - Research Site, Veliko Tarnovo
- Research Site, Mississauga, Ontario, Canada
- Czechia (9):
  - Research Site, Brno
  - Research Site, Bruntál
  - Research Site, Hlučín
  - Research Site, Liberec
  - Research Site, Ostrava
  - Research Site, Ostrava - Poruba
  - Research Site, Ostrava - Trebovice
  - Research Site, Prague
  - Research Site, Zlín
- Germany (3):
  - Research Site, Dresden
  - Research Site, Hamburg
  - Research Site, München
- Hungary (4):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Zalaegerszeg
- Research Site, Amsterdam, Netherlands
- Poland (8):
  - Research Site, Bytom
  - Research Site, Chełm Śląski
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Lodz
  - Research Site, Środa Wielkopolska
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Żyrardów
- Russia (7):
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Petrozavodsk
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Voronezh
  - Research Site, Yaroslavl
- Slovakia (2):
  - Research Site, Trebišov
  - Research Site, Trnava
- South Africa (7):
  - Research Site, Pretoria, Gauteng
  - Research Site, Durban, KwaZulu-Natal
  - Research Site, Cape Town, Western Cape
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Pretoria
  - Research Site, Stellenbosch
- Ukraine (9):
  - Research Site, Donetsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Simferopol
  - Research Site, Zaporyzhzhya
- United Kingdom (8):
  - Research Site, Reading, Berkshire
  - Research Site, London, Greater London
  - Research Site, Eastbourne, Sussex
  - Research Site, Basingstoke
  - Research Site, Eastbourne
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Wolverhampton

REFERENCES:
- [Derived] Taylor PC, Genovese MC, Greenwood M, Ho M, Nasonov E, Oemar B, Stoilov R, Vencovsky J, Weinblatt M. OSKIRA-4: a phase IIb randomised, placebo-controlled study of the efficacy and safety of fostamatinib monotherapy. Ann Rheum Dis. 2015 Dec;74(12):2123-9. doi: 10.1136/annrheumdis-2014-205361. Epub 2014 Jul 29. PMID 25074688

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 452 patients were enrolled into the main study, with 198 patients enrolled into a separate MRI sub-study. Synovitis results for the MRI sub-study were reported later due to study delays and so are presented entirely separately.
Pre-assignment Details: A total of 173 patients failed screening to the main study.
Groups:
- FOSTA 100 MG BID PO: Dosing Group A
- FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO: Dosing Group B
- FOSTA 100 MG BID (4 WKS) THEN 100 MG QD PO: Dosing Group C
- ADALIMUMAB 40 MG SC: Dosing Group D
- PLACEBO (6 WKS) THEN FOSTA 100 MG BID PO: Dosing Group F
- PLACEBO (6 WK) THEN FOSTA 100 MG BID (4 WK) THEN 150 MG QD PO: Dosing Group G
Period: Overall Study
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | FOSTA 100 MG BID (4 WKS) THEN 100 MG QD PO | ADALIMUMAB 40 MG SC | PLACEBO (6 WKS) THEN FOSTA 100 MG BID PO | PLACEBO (6 WK) THEN FOSTA 100 MG BID (4 WK) THEN 150 MG QD PO
Started | 54 (Patients who received treatment) | 48 (Patients who received treatment) | 57 (Patients who received treatment) | 54 (Patients who received treatment) | 27 (Patients who received treatment) | 25 (Patients who received treatment)
Randomised But Did Not Receive Treatment | 2 (Eligibility criteria not fulfilled/subject decision/other) | 5 (Eligibility criteria not fulfilled/subject decision/other) | 2 (Eligibility criteria not fulfilled/subject decision/other) | 3 (Eligibility criteria not fulfilled/subject decision/other) | 2 (Eligibility criteria not fulfilled/subject decision/other) | 0 (Eligibility criteria not fulfilled/subject decision/other)
Completed | 36 (Number of patients who completed treatment includes patients who had a dose reduction.) | 38 (Number of patients who completed treatment includes patients who had a dose reduction.) | 41 (Number of patients who completed treatment includes patients who had a dose reduction.) | 48 (Number of patients who completed treatment includes patients who had a dose reduction.) | 19 (Number of patients who completed treatment includes patients who had a dose reduction.) | 19 (Number of patients who completed treatment includes patients who had a dose reduction.)
Not Completed | 18 | 10 | 16 | 6 | 8 | 6
Not completed — Not reported | 0 | 0 | 1 | 0 | 0 | 0
Not completed — e.g., change in circumstances | 8 | 3 | 3 | 3 | 4 | 4
Not completed — Severe non-compliance to protocol | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Lack of therapeutic response | 1 | 0 | 2 | 1 | 1 | 0
Not completed — Dev. of study specific discont. criteria | 2 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 7 | 7 | 8 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | FOSTA 100 MG BID (4 WKS) THEN 100 MG QD PO | ADALIMUMAB 40 MG SC | PLACEBO (6 WKS) THEN FOSTA 100 MG BID PO | PLACEBO (6 WK) THEN FOSTA 100 MG BID (4 WK) THEN 150 MG QD PO | Total
Number analyzed (Participants) | 54 | 48 | 57 | 54 | 27 | 25 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (11.5) | 50 (12.6) | 50 (11.0) | 48 (12.4) | 50 (12.7) | 53 (10.8) | 50 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 48 | 45 | 20 | 20 | 210
  Male | 16 | 9 | 9 | 9 | 7 | 5 | 55
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 48 | 47 | 48 | 51 | 23 | 23 | 240
  Black or African American | 5 | 0 | 6 | 1 | 3 | 1 | 16
  Asian | 1 | 1 | 0 | 1 | 0 | 1 | 4
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Indian or Pakistani | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Other | 0 | 0 | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: DAS28-CRP Score - Change From Baseline to Week 6 Compared to Placebo
Description: DAS28-CRP: Disease Activity Score based on a count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (CRP) and the patient's own assessment. Scores can take any positive value with a lower value indicating a better clinical condition. Mean changes from baseline in DAS28-CRP score are shown at each visit and are presented as decreases from baseline (defined as baseline minus post-baseline) with larger changes indicative of a better clinical condition. ANCOVA = analysis of covariance, BID = twice daily, CRP = C-reactive protein, DMARD = disease-modifying anti-rheumatic drug, IR = inadequate response, LS = least squares, n/a = not applicable, PO = orally, QD = once a day, SC = subcutaneous.
Time Frame: Baseline and 6 weeks
Population: The full analysis set includes those patients who received at least 1 dose of investigational product. Patients were analysed by randomised treatment in accordance with the intention to treat principle. In line with the study objectives, fostamatinib was compared with placebo (not adalimumab) at Week 6.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Dosing Group A: FOSTA 100 MG BID PO
- Dosing Group B: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO
- Dosing Group C: FOSTA 100 MG BID (4 WKS) THEN 100 MG QD PO
- Dosing Group E: PLACEBO (COMBINED)
Arm/Group | Dosing Group A | Dosing Group B | Dosing Group C | Dosing Group E
Number analyzed (Participants) | 54 | 48 | 57 | 52
Units on a scale | 1.1 (0.92) [lower limit 0.23] | 1.1 (1.01) | 0.8 (0.96) | 0.6 (1.14)
Statistical Analysis 1: Comparison: Dosing Group A vs Dosing Group E; Change from baseline at Week 6. Non-responder imputation applied following premature withdrawal, or any DMARD initiation, or for 8 weeks following receipt of parenteral steroids, or for patients with no post baseline data; Test type: Superiority or Other; p = 0.006, ANCOVA; Includes terms for baseline as a continuous covariate and treatment, DMARD naivety (DMARD naive vs DMARD-IR/intolerant) and pooled country as factors; Treatment difference = 0.56, 90% CI 2-sided [0.23 to 0.90]
Statistical Analysis 2: Comparison: Dosing Group B vs Dosing Group E; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.022, ANCOVA; [statistical method as in outcome 1, analysis 1]; Treatment difference = 0.49, 90% CI 2-sided [0.14 to 0.84]
Statistical Analysis 3: Comparison: Dosing Group C vs Dosing Group E; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.280, ANCOVA; [statistical method as in outcome 1, analysis 1]; Treatment difference = 0.22, 90% CI 2-sided [-0.12 to 0.56]

2. Primary Outcome: DAS28-CRP Score - Change From Baseline to Week 24 Compared to Adalimumab
Description: DAS28-CRP: Disease Activity Score based on a count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (CRP) and the patient's own assessment. Scores can take any positive value with a lower value indicating a better clinical condition. Mean changes from baseline in DAS28-CRP score are shown at each visit and are presented as decreases from baseline (defined as baseline minus post-baseline) with larger changes indicative of a better clinical condition. Non-responder imputation has been applied by carrying the baseline observation forward. ANCOVA = analysis of covariance, BID = twice daily, CRP = C-reactive protein, DMARD = disease-modifying anti-rheumatic drug, IR = inadequate response, LS = least squares, n/a = not applicable, PO = orally, QD = once a day, SC = subcutaneous.
Time Frame: Baseline and 24 weeks
Population: The full analysis set includes those patients who received at least 1 dose of investigational product. Patients were analysed by randomised treatment in accordance with the intention to treat principle. In line with the study objectives, fostamatinib was compared with adalimumab (not placebo) at Week 24.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Dosing Group D: ADALIMUMAB 40 MG SC
- Dosing Group F: PLACEBO (6 WKS) THEN FOSTA 100 MG BID PO
- Dosing Group G: PLACEBO (6 WK) THEN FOSTA 100 MG BID (4 WK) THEN 150 MG QD PO
Arm/Group | Dosing Group A | Dosing Group B | Dosing Group C | Dosing Group D | Dosing Group F | Dosing Group G
Number analyzed (Participants) | 54 | 48 | 57 | 54 | 27 | 25
Units on a scale | 1.0 (1.31) | 1.1 (1.22) | 1.0 (1.25) | 1.8 (1.45) | 1.1 (1.26) | 1.4 (1.26)
Statistical Analysis 1: Comparison: Dosing Group A vs Dosing Group D; Change from baseline at Week 24. Non-responder imputation applied following premature withdrawal, or any DMARD initiation, or for 8 weeks following receipt of parenteral steroids, or for patients with no post baseline data; Test type: Non-Inferiority or Equivalence — For the comparison with adalimumab a non-inferiority margin of -0.6 in the mean change from baseline in DAS28-CRP at Week 24 was defined. The lower 80% confidence interval for treatment difference was below this value so non-inferiority could not be concluded. A p-value is also provided for a 2-sided test of superiority; p = 0.005, ANCOVA; [statistical method as in outcome 1, analysis 1]; Treatment difference = -0.72, 80% CI 2-sided [-1.04 to -0.40]
Statistical Analysis 2: Comparison: Dosing Group B vs Dosing Group D; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.020, ANCOVA; [statistical method as in outcome 1, analysis 1]; Treatment difference = -0.61, 80% CI 2-sided [-0.94 to -0.27]
Statistical Analysis 3: Comparison: Dosing Group C vs Dosing Group D; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.004, ANCOVA; [statistical method as in outcome 1, analysis 1]; Treatment difference = -0.72, 80% CI 2-sided [-1.04 to -0.40]

3. Secondary Outcome: DAS28 EULAR Response at Week 6
Description: Change in DAS28 was derived for each post baseline scheduled assessment and categorised using the European League Against Rheumatism (EULAR) response criteria. Non-responder imputation has been applied by carrying the baseline observation forward. bid = twice daily, DAS28 = Disease Activity Score based on a 28-joint count, DMARD = disease-modifying anti-rheumatic drug, OR = odds ratio, PO = orally, qd = once a day, SC = subcutaneous.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | Dosing Group A | Dosing Group B | Dosing Group C | Dosing Group D | Dosing Group E
Number analyzed (Participants) | 54 | 48 | 57 | 54 | 52
Percentage of responders
  No response | 37.0 (1.46) [0.20 to 0.68] | 33.3 (1.34) [0.26 to 0.89] | 57.9 (1.30) [0.20 to 0.65] | 40.7 (1.58) | 67.3 (1.33)
  Moderate response | 53.7 | 47.9 | 35.1 | 38.9 | 25.0
  Good response | 9.3 | 18.8 | 7.0 | 20.4 | 7.7
Statistical Analysis 1: Comparison: Dosing Group A vs Dosing Group E; Non-responder imputation has been applied following premature withdrawal, or any DMARD initiation, or for 8 weeks following receipt of any parenteral steroids, or for patients with no post baseline data; Test type: Superiority or Other; p = 0.005, Proportional odds model; Odds Ratio (OR) = 3.05, 90% CI 2-sided [1.59 to 5.86] — An odds ratio >1 indicates a benefit towards fostamatinib
Statistical Analysis 2: Comparison: Dosing Group B vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Proportional odds model; Odds Ratio (OR) = 4.11, 90% CI 2-sided [2.10 to 8.05] — An odds ratio >1 indicates a benefit towards fostamatinib
Statistical Analysis 3: Comparison: Dosing Group C vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.335, Proportional odds model; Odds Ratio (OR) = 1.47, 90% CI 2-sided [0.76 to 2.83] — An odds ratio >1 indicates a benefit towards fostamatinib

4. Secondary Outcome: DAS28 EULAR Response at Week 24
Description: as for outcome 3
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of responders
Arm/Group | Dosing Group A | Dosing Group B | Dosing Group C | Dosing Group D | Dosing Group F | Dosing Group G
Number analyzed (Participants) | 54 | 48 | 57 | 54 | 27 | 25
Percentage of responders
  No response | 51.9 (1.46) [0.20 to 0.68] | 41.7 (1.34) [0.26 to 0.89] | 52.6 (1.30) [0.20 to 0.65] | 31.5 (1.58) | 55.6 (1.33) | 40.0 (1.48)
  Moderate response | 29.6 | 39.6 | 29.8 | 27.8 | 33.3 | 36.0
  Good response | 18.5 | 18.8 | 17.5 | 40.7 | 11.1 | 24.0
Statistical Analysis 1: Comparison: Dosing Group A vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.007, Proportional odds model; Odds Ratio (OR) = 0.37, 90% CI 2-sided [0.20 to 0.68] — An odds ratio >1 indicates a benefit towards fostamatinib
Statistical Analysis 2: Comparison: Dosing Group B vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.051, Proportional odds model; Odds Ratio (OR) = 0.48, 90% CI 2-sided [0.26 to 0.89] — An odds ratio >1 indicates a benefit towards fostamatinib
Statistical Analysis 3: Comparison: Dosing Group C vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.004, Proportional odds model; Odds Ratio (OR) = 0.36, 90% CI 2-sided [0.20 to 0.65] — An odds ratio >1 indicates a benefit towards fostamatinib

5. Secondary Outcome: Proportion of Patients Achieving ACR20 up to Week 24
Description: ACR20: American College of Rheumatology 20% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as CRP) and the physician and patient's own assessments of disease activity, pain and physical function. Non-responder imputation has been applied by carrying the baseline observation forward. BID = twice daily, CRP = C-reactive protein, DMARD = disease-modifying anti-rheumatic drug, IR = inadequate response, n/a = not applicable, PO = orally, qd = once a day, SC = subcutaneous.
Time Frame: 6 and 24 weeks
Population: The full analysis set includes those patients who received at least 1 dose of investigational product. Patients were analysed by randomised treatment in accordance with the intention to treat principle. In line with the study objectives, fostamatinib was compared with placebo (not adalimumab) at Week 6 and with adalimumab (not placebo) at Week 24.
Measure: Number; unit: Percentage of responders
Arm/Group | Dosing Group A | Dosing Group B | Dosing Group C | Dosing Group D | Dosing Group E | Dosing Group F | Dosing Group G
Number analyzed (Participants) | 54 | 48 | 57 | 54 | 52 | 27 | 25
Percentage of responders
  Week 6 | 48.1 | 47.9 | 38.6 | 53.7 | 19.2 | NA — Data appears under Group E at Week 6. | NA — Data appears under Group E at Week 6.
  Week 24 | 40.7 | 56.3 | 35.1 | 59.3 | NA — Data appears under Groups F and G at Week 24. | 44.4 | 44.0
Statistical Analysis 1: Comparison: Dosing Group A vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mantel Haenszel — Week 6; p-values are calculated using a Mantel-Haenszel approach stratified by DMARD naivety (DMARD naive vs DMARD-IR/intolerant) and pooled country; Weighted difference in proportions = 0.29, 90% CI 2-sided [0.17 to 0.40] — 90% confidence intervals are calculated using a Mantel-Haenszel approach stratified by DMARD naivety (DMARD naive vs DMARD-IR/intolerant) and pooled country
Statistical Analysis 2: Comparison: Dosing Group B vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mantel Haenszel — Week 6; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = 0.30, 90% CI 2-sided [0.18 to 0.43] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Dosing Group C vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.007, Mantel Haenszel — Week 6; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = 0.19, 90% CI 2-sided [0.07 to 0.31] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Dosing Group A vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.049, Mantel Haenszel — Week 24; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = -0.16, 90% CI 2-sided [-0.30 to -0.03] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Dosing Group B vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.803, Mantel Haenszel — Week 24; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = -0.02, 90% CI 2-sided [-0.16 to 0.12] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Dosing Group C vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.003, Mantel Haenszel — Week 24; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = -0.24, 90% CI 2-sided [-0.37 to -0.10] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Proportion of Patients Achieving ACR50 up to Week 24
Description: ACR50: American College of Rheumatology 50% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as CRP) and the physician and patient's own assessments of disease activity, pain and physical function. Non-responder imputation has been applied by carrying the baseline observation forward. BID = twice daily, CRP = C-reactive protein, DMARD = disease-modifying anti-rheumatic drug, IR = inadequate response, n/a = not applicable, PO = orally, qd = once a day, SC = subcutaneous.
Time Frame: 6 and 24 weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of responders
Arm/Group | Dosing Group A | Dosing Group B | Dosing Group C | Dosing Group D | Dosing Group E | Dosing Group F | Dosing Group G
Number analyzed (Participants) | 54 | 48 | 57 | 54 | 52 | 27 | 25
Percentage of responders
  Week 6 | 13.0 | 12.5 | 7.0 | 25.9 | 3.8 | NA — Data appears under Group E at Week 6. | NA — Data appears under Group E at Week 6.
  Week 24 | 20.4 | 18.8 | 12.3 | 31.5 | NA — Data appears under Groups F and G at Week 24. | 22.2 | 24.0
Statistical Analysis 1: Comparison: Dosing Group A vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.059, Mantel Haenszel — Week 6; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = 0.09, 90% CI 2-sided [0.01 to 0.18] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Dosing Group B vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.071, Mantel Haenszel — Week 6; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = 0.09, 90% CI 2-sided [0.01 to 0.17] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Dosing Group C vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.758, Mantel Haenszel — Week 6; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = 0.01, 90% CI 2-sided [-0.05 to 0.07] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Dosing Group A vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.114, Mantel Haenszel — Week 24; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = -0.12, 90% CI 2-sided [-0.24 to 0.00] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Dosing Group B vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.078, Mantel Haenszel — Week 24; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = -0.14, 90% CI 2-sided [-0.26 to -0.01] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Dosing Group C vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.003, Mantel Haenszel — Week 24; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = -0.21, 90% CI 2-sided [-0.32 to -0.09] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Proportion of Patients Achieving ACR70 up to Week 24
Description: ACR70: American College of Rheumatology 70% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as CRP) and the physician and patient's own assessments of disease activity, pain and physical function. Non-responder imputation has been applied by carrying the baseline observation forward. BID = twice daily, CRP = C-reactive protein, DMARD = disease-modifying anti-rheumatic drug, IR = inadequate response, n/a = not applicable, PO = orally, qd = once a day, SC = subcutaneous.
Time Frame: 6 and 24 weeks
Population: as for outcome 5
Measure: Number; unit: Percentage of responders
Arm/Group | Dosing Group A | Dosing Group B | Dosing Group C | Dosing Group D | Dosing Group E | Dosing Group F | Dosing Group G
Number analyzed (Participants) | 54 | 48 | 57 | 54 | 52 | 27 | 25
Percentage of responders
  Week 6 | 1.9 | 4.2 | 1.8 | 7.4 | 3.8 | NA — Data appears under Group E at Week 6. | NA — Data appears under Group E at Week 6.
  Week 24 | 9.3 | 10.4 | 3.5 | 20.4 | NA — Data appears under Groups F and G at Week 24. | 7.4 | 4.0
Statistical Analysis 1: Comparison: Dosing Group A vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.460, Mantel Haenszel — Week 6; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = -0.02, 90% CI 2-sided [-0.07 to 0.03] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Dosing Group B vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.903, Mantel Haenszel — Week 6; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = 0.00, 90% CI 2-sided [-0.05 to 0.06] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Dosing Group C vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.172, Mantel Haenszel — Week 6; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = -0.03, 90% CI 2-sided [-0.08 to 0.01] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Dosing Group A vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.082, Mantel Haenszel — Week 24; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = -0.11, 90% CI 2-sided [-0.21 to -0.01] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Dosing Group B vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.092, Mantel Haenszel — Week 24; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = -0.11, 90% CI 2-sided [-0.21 to -0.00] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Dosing Group C vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.002, Mantel Haenszel — Week 24; [statistical method as in outcome 5, analysis 1]; Weighted difference in proportions = -0.17, 90% CI 2-sided [-0.27 to -0.08] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: ACRn - Comparison Between Fostamatinib and Placebo at Week 6
Description: ACRn: American College of Rheumatology Index of RA improvement, based on smallest percentage improvement in the count of swollen joints (out of 28 joints), count of tender joints (out of 28 joints) or in blood test measures of inflammation (such as CRP) or the physician and patient's own asessment of disease activity, pain and physical function. Scores are reported as a percentage improvement on a scale of -100 to +100, with larger values representing a better clinical outcome. Non-responder imputation has been applied by carrying the baseline observation forward. BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, IR = inadequate response, n/a = not applicable, PO = orally, qd = once a day, SC = subcutaneous. Mean refers to change at Week 6. Treatment difference: difference between fostamatinib and placebo groups.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage improvement from baseline
Arm/Group | Dosing Group A | Dosing Group B | Dosing Group C | Dosing Group D | Dosing Group E
Number analyzed (Participants) | 54 | 48 | 57 | 54 | 52
Percentage improvement from baseline | 16.60 (30.682) | 15.07 (33.334) | 6.48 (32.237) | 15.53 (43.015) | -6.49 (35.159)
Statistical Analysis 1: Comparison: Dosing Group A vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Van Elteren; Estimated using the Van Elteren test stratified by DMARD naivety (DMARD naive vs DMARD-IR/intolerant) and pooled country; Treatment difference = 23.39, 90% CI 2-sided [9.57 to 40.00]
Statistical Analysis 2: Comparison: Dosing Group B vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.006, Van Elteren; [statistical method as in outcome 8, analysis 1]; Treatment difference = 22.97, 90% CI 2-sided [7.84 to 38.34]
Statistical Analysis 3: Comparison: Dosing Group C vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.234, Van Elteren; [statistical method as in outcome 8, analysis 1]; Treatment difference = 5.72, 90% CI 2-sided [-3.20 to 21.68]

9. Secondary Outcome: ACRn - Comparison Between Fostamatinib and Adalimumab at Week 24
Description: ACRn: American College of Rheumatology Index of RA improvement, based on smallest percentage improvement in the count of swollen joints (out of 28 joints), count of tender joints (out of 28 joints) or in blood test measures of inflammation (such as CRP) or the physician and patient's own asessment of disease activity, pain and physical function. Scores are reported as a percentage improvement on a scale of -100 to +100, with larger values representing a better clinical outcome. Non-responder imputation has been applied by carrying the baseline observation forward. BID = twice daily, CRP = C-reactive protein, DMARD = disease-modifying anti-rheumatic drug, IR = inadequate response, n/a = not applicable, PO = orally, qd = once a day, SC = subcutaneous. Mean refers to change at Week 24. Treatment difference: difference between fostamatinib and adalimumab groups.
Time Frame: Baseline and 24 weeks
Population: The full analysis set includes those patients who received at least 1 dose of investigational product. Patients were analysed by randomised treatment in accordance with the intention to treat principle.In line with the study objectives, fostamatinib was compared with adalimumab (not placebo) at Week 24.
Measure: Mean (Standard Deviation); unit: Percentage improvement from baseline
Arm/Group | Dosing Group A | Dosing Group B | Dosing Group C | Dosing Group D
Number analyzed (Participants) | 54 | 48 | 57 | 54
Percentage improvement from baseline | 18.35 (34.355) | 22.03 (32.361) | 11.49 (26.916) | 31.21 (39.187)
Statistical Analysis 1: Comparison: Dosing Group A vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.030, Van Elteren; [statistical method as in outcome 8, analysis 1]; Treatment difference = -13.72, 90% CI 2-sided [-25.01 to 0.00]
Statistical Analysis 2: Comparison: Dosing Group B vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.207, Van Elteren; [statistical method as in outcome 8, analysis 1]; Treatment difference = -9.49, 90% CI 2-sided [-25.00 to 6.96]
Statistical Analysis 3: Comparison: Dosing Group C vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.002, Van Elteren; [statistical method as in outcome 8, analysis 1]; Treatment difference = -19.53, 90% CI 2-sided [-30.01 to -6.25]

10. Secondary Outcome: HAQ-DI - Comparison of the Change From Baseline Between Fostamatinib and Placebo at Week 6
Description: HAQ-DI: Health Assessment Questionnaire - Disability Index, a measure of physical function. The HAQ-DI score is calculated by summing the category scores from 8 sub-categories (ie, scores for patient ability in dressing and grooming, rising, eating, walking, hygiene, reach, grip and common daily activities) and dividing by the number of categories completed. The HAQ-DI score takes values between 0 and 3, with a higher score indicating greater disability. Non-responder imputation has been applied by carrying the baseline observation forward. ANCOVA = analysis of covariance, BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, IR = inadequate response, LS = least squares, n/a = not applicable, PO = orally, qd = once a day, SC = subcutaneous.
Time Frame: Baseline and 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dosing Group A | Dosing Group B | Dosing Group C | Dosing Group D | Dosing Group E
Number analyzed (Participants) | 54 | 48 | 57 | 54 | 52
Units on a scale | 0.3 (0.35) | 0.3 (0.54) | 0.2 (0.43) | 0.3 (0.45) | 0.1 (0.52)
Statistical Analysis 1: Comparison: Dosing Group A vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.007, ANCOVA; Including terms for baseline as a continuous covariate & treatment, DMARD naivety (DMARD naive vs DMARD-IR/intolerant) & pooled country as factors; Treatment difference = 0.24, 90% CI 2-sided [0.09 to 0.38]
Statistical Analysis 2: Comparison: Dosing Group B vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.016, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment difference = 0.22, 90% CI 2-sided [0.07 to 0.37]
Statistical Analysis 3: Comparison: Dosing Group C vs Dosing Group E; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.094, ANCOVA; Includes terms for baseline as a continuous covariate & treatment, DMARD naivety (DMARD naive vs DMARD-IR/intolerant) & pooled country as factors; Treatment difference = 0.14, 90% CI 2-sided [0.00 to 0.29]

11. Secondary Outcome: HAQ-DI - Comparison of the Change From Baseline Between Fostamatinib and Adalimumab at Week 24
Description: as for outcome 10
Time Frame: Baseline and 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dosing Group A | Dosing Group B | Dosing Group C | Dosing Group D | Dosing Group F | Dosing Group G
Number analyzed (Participants) | 54 | 48 | 57 | 54 | 27 | 25
Units on a scale | 0.3 (0.57) | 0.4 (0.56) | 0.2 (0.45) | 0.5 (0.53) | 0.3 (0.47) | 0.1 (0.35)
Statistical Analysis 1: Comparison: Dosing Group A vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.043, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment difference = -0.20, 90% CI 2-sided [-0.36 to -0.04]
Statistical Analysis 2: Comparison: Dosing Group B vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.158, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment difference = -0.14, 90% CI 2-sided [-0.31 to 0.02]
Statistical Analysis 3: Comparison: Dosing Group C vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.001, ANCOVA; [statistical method as in outcome 10, analysis 3]; Treatment difference = -0.32, 90% CI 2-sided [-0.47 to -0.16]

12. Secondary Outcome: SF-36 - Comparison of the Change in PCS From Baseline Between Fostamatinib and Adalimumab at Week 24
Description: SF-36: 36-item Short Form Health Survey, a measure of health-related QoL. Scores for 8 sub-domains (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Function, Role-Emotional & Mental Health) are derived & normalised to a scale of 0-100. Physical & Mental Component Scores (PCS & MCS) are derived by multiplying each of these 8 scores by a constant, summing them & standardising against a population with mean of 50, standard deviation of 10. Higher scores represent a better QoL. Mean changes from baseline score are presented at each visit as increases from baseline (defined as post-baseline minus baseline); larger changes indicate a better clinical condition. Non-responder imputation applied by carrying the baseline observation forward. ANCOVA = analysis of covariance, BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, IR = inadequate response, LS = least squares, PO = orally, QD = once a day, QoL = quality of life, SC = subcutaneous.
Time Frame: Baseline and 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dosing Group A | Dosing Group B | Dosing Group C | Dosing Group D | Dosing Group F | Dosing Group G
Number analyzed (Participants) | 54 | 48 | 57 | 54 | 27 | 25
Units on a scale | 4 (7.3) | 5 (7.2) | 4 (7.4) | 7 (8.4) | 4 (8.7) | 3 (5.0)
Statistical Analysis 1: Comparison: Dosing Group A vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.050, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment difference = -2.77, 90% CI 2-sided [-5.08 to -0.45]
Statistical Analysis 2: Comparison: Dosing Group B vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.360, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment difference = -1.33, 90% CI 2-sided [-3.73 to 1.06]
Statistical Analysis 3: Comparison: Dosing Group C vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.032, ANCOVA; [statistical method as in outcome 10, analysis 3]; Treatment difference = -2.99, 90% CI 2-sided [-5.29 to -0.70]

13. Secondary Outcome: SF-36 - Comparison of the Change in MCS From Baseline Between Fostamatinib and Adalimumab at Week 24
Description: as for outcome 12
Time Frame: Baseline and 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dosing Group A | Dosing Group B | Dosing Group C | Dosing Group D | Dosing Group F | Dosing Group G
Number analyzed (Participants) | 54 | 48 | 57 | 54 | 27 | 25
Units on a scale | 3 (9.3) | 3 (11.5) | 2 (10.0) | 4 (9.8) | 3 (5.9) | 0 (10.1)
Statistical Analysis 1: Comparison: Dosing Group A vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.568, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment difference = -1.02, 90% CI 2-sided [-3.95 to 1.92]
Statistical Analysis 2: Comparison: Dosing Group B vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.368, ANCOVA; [statistical method as in outcome 10, analysis 1]; Treatment difference = -1.66, 90% CI 2-sided [-4.69 to 1.38]
Statistical Analysis 3: Comparison: Dosing Group C vs Dosing Group D; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.160, ANCOVA; [statistical method as in outcome 10, analysis 3]; Treatment difference = -2.48, 90% CI 2-sided [-5.38 to 0.43]

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: For placebo treated patients time frame includes both placebo(6 weeks) and fostamatinib(18 weeks) treatment. 1 SAE occurred in these treatment arms began during the 6 week placebo treated period
Groups:
- ADALIMUMAB 40 MG: Dosing Group D
- FOSTA 100 MG BID: Dosing Group A
- FOSTA 100 MG BID (4 WKS) THEN 100 MG QD: Dosing Group C
Arm/Group | ADALIMUMAB 40 MG | FOSTA 100 MG BID | FOSTA 100 MG BID (4 WKS) THEN 100 MG QD | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD | PLACEBO (6 WKS) FOSTA 100 MG BID (4 WKS) 150 MG QD-FOSTAperiod | PLACEBO (6 WKS) FOSTA 100 MG BID (4 WKS) 150 MG QD-PBO Period | PLACEBO (6 WKS) THEN FOSTA 100 MG BID - FOSTA Period | PLACEBO (6 WKS) THEN FOSTA 100 MG BID - Placebo Period
Serious Adverse Events (participants affected / at risk) | 4/54 | 5/54 | 4/57 | 1/48 | 0/25 | 1/25 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 15/54 | 30/54 | 19/57 | 20/48 | 13/25 | 1/25 | 11/27 | 3/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADALIMUMAB 40 MG (N=54) | FOSTA 100 MG BID (N=54) | FOSTA 100 MG BID (4 WKS) THEN 100 MG QD (N=57) | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD (N=48) | PLACEBO (6 WKS) FOSTA 100 MG BID (4 WKS) 150 MG QD-FOSTAperiod (N=25) | PLACEBO (6 WKS) FOSTA 100 MG BID (4 WKS) 150 MG QD-PBO Period (N=25) | PLACEBO (6 WKS) THEN FOSTA 100 MG BID - FOSTA Period (N=27) | PLACEBO (6 WKS) THEN FOSTA 100 MG BID - Placebo Period (N=27)
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COR PULMONALE ACUTE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERADRENALISM (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHRONIC SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS CHRONIC (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENISCUS LESION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC MYXOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ESSENTIAL HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADALIMUMAB 40 MG (N=54) | FOSTA 100 MG BID (N=54) | FOSTA 100 MG BID (4 WKS) THEN 100 MG QD (N=57) | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD (N=48) | PLACEBO (6 WKS) FOSTA 100 MG BID (4 WKS) 150 MG QD-FOSTAperiod (N=25) | PLACEBO (6 WKS) FOSTA 100 MG BID (4 WKS) 150 MG QD-PBO Period (N=25) | PLACEBO (6 WKS) THEN FOSTA 100 MG BID - FOSTA Period (N=27) | PLACEBO (6 WKS) THEN FOSTA 100 MG BID - Placebo Period (N=27)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 9 (9) | 12 (12) | 13 (13) | 4 (4) | 0 (0) | 3 (3) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
NASOPHARYNGITIS (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 5 (5) | 7 (7) | 5 (5) | 3 (3) | 7 (7) | 0 (0) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor can review and comment on results communications prior to publication. Sponsor will be allowed a review period of at least 60 days from submission but can request that publication be delayed for a period up to 6 months. Any reasonable comments made by the sponsor will be incorporated by the PI into the publication.